CLINICAL TRIAL: NCT04866316
Title: Protocol for a Mixed Methods and Multi-site Assessment of the Implementation Process and Outcomes of a New Community-based Frailty Programme
Brief Title: Protocol for Multi-site Evaluation of New Community-based Frailty Programme
Status: Completed | Type: Observational
Sponsor: Geriatric Education and Research Institute (Other Government)
Collaborators: Alexandra Hospital (Other); Changi General Hospital (Other); Ng Teng Fong General Hospital (Other); Sengkang General Hospital (Other); Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/00925
Record Dates: First submitted 2021-04-12; First posted 2021-04-29 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-08

CONDITIONS: Frailty; Frail Elderly Syndrome; Frailty Syndrome
Keywords: frailty care; comprehensive geriatric assessment; care coordination; multidisciplinary team care
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GSH Participants: Qualitative - Semi-structured focus group discussions with care recipients
  Quantitative - Pre-test post-test design using survey-based data collection
  Quantitative - Retrospective cohort design with propensity score matched comparators
  Interventions: Other: There is no active intervention as this is a service evaluation
- Policy owners, implementers & care partners, health and social care professionals: Qualitative - Semi-structured in-depth interview with key policy and programme decision-makers
  Qualitative - Semi-structured focus group discussions with health and social care professionals
  Qualitative - Participant observations
  Quantitative - Longitudinal monitoring of process indicators
  Interventions: Other: There is no active intervention as this is a service evaluation

INTERVENTIONS:
Other: There is no active intervention as this is a service evaluation — There is no active intervention as this is a service evaluation

SUMMARY:
Background: Frailty is increasing in prevalence internationally with population ageing. Frailty can be managed or even reversed through community-based interventions delivered by a multi-disciplinary team of professionals, but to varying degrees of effectiveness. However, many of the implementation insights of these care models are contextual, and may not be applicable in different cultural contexts. The Geriatric Service Hub (GSH) is a novel frailty care programme in Singapore, that includes key components of frailty care such as comprehensive geriatric assessments, care coordination and the assembly of a multidisciplinary team. The aim of this study is to gain insights on the factors influencing the implementation approaches adopted by five participating sites, and the effectiveness of the programme.

Methods: We will adopt a mixed-methods approach that includes a qualitative evaluation among key stakeholders and participants taking part in the programme, through in depth-interviews and focus group discussions. The main topics covered includes factors that affected the development and implementation of each programme, operations and other contextual factors that influenced implementation outcomes. The quantitative evaluation (1) monitors each programme's care process through quality indicators, (2) a multiple-time point survey study to compare programme participants' pre- and post- outcomes on patient engagement (collaboRATE and 13-item Patient Activation Measure;PAM), healthcare experiences (Consumer Assessment of Healthcare Providers and System Clinician and Group Survey Version 3.0; CG-CAHPS), health status and quality of life (Barthel Index of Activities of Daily Living, fall counts, the EuroQol questionnaire and the Control, Autonomy, Self-realization and Pleasure scale; CASP-19), impact on caregivers (Zarit Burden Interview) and societal costs (Client Service Receipt Inventory). (3) A retrospective cohort design to assess healthcare and cost utilisation between participants of the programme and a propensity score matched comparator group.

Discussion: The GSH sites share a common goal to increasing accessibility of essential services to frail older adults, and providing comprehensive care. The results of this evaluation study will provide valuable evidence to the impact and effectiveness of the GSH, and inform to the design of similar programmes targeting frail older adults.

ELIGIBILITY:
1. Qualitative In depth Interviews/ Policy owners & administrators

   Inclusion Criteria:
   * Decision-makers who are higher-level administrators or clinicians who have the authority to make policy and implementation decisions and/ or
   * Individuals who are familiar with the hospital's overall frailty strategy; and/ or
   * Individuals that who led the development and implementation of the programme

   Exclusion Criteria:
   * Do not meet inclusion criteria above
2. Qualitative Focus group discussions/ Implementation team

   Inclusion Criteria:
   * Individuals with time funded through the programme who have been providing services in the GSH for at least six month

   Exclusion Criteria:
   * Do not meet inclusion criteria above
3. Qualitative Focus group discussions/ partner organizations

   Inclusion Criteria:
   * healthcare professionals and administrative staff who provided services within the new programme for at least six months

   Exclusion Criteria:
   * Do not meet inclusion criteria above
4. Qualitative Focus group discussions/ GSH participants

   Inclusion Criteria:
   * Participants who receive care under the new model for at least three months

   Exclusion Criteria:
   * Do not meet inclusion criteria above
5. Quantitative survey questionnaire / GSH participants

Inclusion Criteria:

* Patients that meet the necessary clinical criteria for enrollment in the respective GSH programme
* Age: 65 and above
* Clinical Frailty Score (CFS): 4-7

Exclusion Criteria:

* Do not meet inclusion criteria above

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Given that the study involves a mixed method evaluation evaluation methodology, to gain a comprehensive understanding of the factors influencing the effectiveness of the implementation approaches adopted by the GSH programmes, and their impacts, the study population will comprise of professional stakeholders playing critical roles in the development and implementation of the new model of community-based frailty care, and the participants of the GSH programme services .
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Functional status | April 2019 - September 2022
  It is hypothesised that better functional status, might reduce the healthcare utilisation (emergency hospitalisation, nursing home admission), caregiver burden and the associated indirect cost. In turn, we might expect overall costs to be lower compared to the comparison group.
  Changes in functional status will be measured using the Barthel Index of Activities of Daily Living (ADL) and Count of falls questionnaire.
Health outcomes | April 2019 - September 2022
  It is hypothesised that better health outcomes, might reduce the healthcare utilisation (emergency hospitalisation, nursing home admission), caregiver burden and the associated indirect cost. In turn, we might expect overall costs to be lower compared to the comparison group.
  Health outcomes will be measured using Quality of Life Questionnaire (EuroQol-5D-5L) and 19-item Quality of Life Scale (CASP-19).

SECONDARY OUTCOMES:
Utilisation of appropriate services | April 2019 - September 2022
  GSH sites offer a range of medical, social and other services through either direct provision or referrals. Given that the model is intended to bridge service gaps (conduct of Comprehensive Geriatric Assessment/ CGA in the community), in the short-term, we hypothesis an increase in the utilisation of appropriate services (rehabilitation, ambulatory services) in this time-limited programme.
  Utilisation of services will be measured using Client Service Receipt Inventory (CSRI).
Patient Satisfaction | April 2019 - September 2022
  GSH participants are expected to benefit from the comprehensive package of health and social services and multidisciplinary team approach. With better care coordination and improved access, it is likely to elicit a higher level of satisfaction relative to comparator groups.
  Patient satisfaction will be measured using the Consumer Assessment of Healthcare Providers and System Clinician & Group Survey Version 3.0 (CG-CAHPS) tool.
Shared decision making/ engagement | April 2019 - September 2022
  Education of the client about self-care, and making decisions about potential care options with inputs from a multidisciplinary team, is expected to result in higher level of shared decision making and engagement relative to comparator groups.
  Shared decision making/ engagement will be measured using the collaboRATE For Patient - 5-point anchor scale, and 13-item Patient Activation Measure (PAM-13).

CONTACTS AND LOCATIONS:
Overall Officials: Woan Shin Tan, PhD, Principal Investigator — Joint Faculty and PI
Locations (1):
- Geriatric Education and Research Institite, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
The information will not be shared due to confidentiality

REFERENCES:
- [Derived] Tan WS, Nai ZL, Tan HTR, Nicholas S, Choo R, Ginting ML, Tan E, Teng PHJ, Lim WS, Wong CH, Ding YY; Geriatric Services Hub Programme Group. Protocol for a mixed-methods and multi-site assessment of the implementation process and outcomes of a new community-based frailty programme. BMC Geriatr. 2022 Jul 15;22(1):586. doi: 10.1186/s12877-022-03254-6. PMID 35840898

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT04866316/Prot_SAP_000.pdf